CLINICAL TRIAL: NCT04656561
Title: A Phase 2, Multicenter, Randomized, Parallel-Group, Double-Masked, 4-Arm, Sham-Controlled Study of the Efficacy, Safety, and Tolerability of ANX007 Administered by Intravitreal Injection in Patients With Geographic Atrophy (GA) Secondary to Age-Related Macular Degeneration (AMD) - The ARCHER Study
Brief Title: A Study Investigating the Efficacy and Safety of Intravitreal Injections of ANX007 in Patients With Geographic Atrophy
Acronym: ARCHER
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Annexon, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ANX007-GA-01
Record Dates: First submitted 2020-12-01; First posted 2020-12-07 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Geographic Atrophy
MeSH Terms: conditions — Geographic Atrophy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- ANX007 Group 1 (Experimental): ANX007 administered every month
  Interventions: Drug: ANX007
- ANX007 Group 2 (Experimental): ANX007 administered every other month
  Interventions: Drug: ANX007
- Sham Group 3 (Sham Comparator): Sham injection administered every month
  Interventions: Other: Sham comparator
- Sham Group 4 (Sham Comparator): Sham injection administered every other month
  Interventions: Other: Sham comparator

INTERVENTIONS:
Drug: ANX007 — Form: solution for injection; Route of Administration: IVT
  Arms: ANX007 Group 1; ANX007 Group 2
Other: Sham comparator — Form and Route of Administration: pressure to mimic IVT injection
  Arms: Sham Group 3; Sham Group 4

SUMMARY:
This study is being conducted in participants with geographic atrophy (GA) secondary to age-related macular degeneration (AMD) to determine if intravitreal (IVT) injections of ANX007 reduce GA lesion growth rate. The results will be used to guide further development of ANX007 in participants with geographic atrophy. The total duration of participation is expected to be approximately 19 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of geographic atrophy of the macula secondary to age-related macular degeneration as determined by the Investigator and confirmed by the Central Reading Center.
* GA lesion must have the following characteristics as determined by the independent Central Reading Center based on assessment of FAF imaging at screening:

  1. Well-demarcated GA with a total area (baseline lesion size) ≥2.5 millimeter squared (mm^2) and ≤17.5 mm^2.
  2. If GA is multifocal, at least 1 focal lesion must measure ≥1.25 mm^2 with the overall aggregate area of GA as specified above.
  3. Presence of hyper autofluorescence, any pattern, in the junctional zone of the GA. Absence of hyper autofluorescence (that is, pattern = none) is exclusionary.
  4. The entire GA lesion must be completely visualized on the macula centered image and must be able to be imaged in its entirety and not contiguous with any peripapillary atrophy.
* Normal luminance BCVA of 24 to 83 letters, inclusive, using ETDRS charts (20/25 to 20/320 Snellen equivalent, inclusive).
* A female participant is eligible if she is not pregnant or breastfeeding and is a woman of non-childbearing potential or is using a contraceptive method that is highly effective, with a failure rate of <1% during the study intervention period and for at least 30 days after the last dose of study intervention.

Exclusion Criteria:

* Geographic atrophy due to other causes than AMD such as Stargardt disease, cone-rod dystrophy, pathologic myopia, or toxic maculopathies (for example, plaquenil maculopathy) in either eye.
* Any evidence of choroidal neovascularization (CNV) in the study eye:

  1. Any history of CNV of any cause based on medical history.
  2. Evidence of prior or active CNV or related findings (for example, retinal pigment epithelial rips or tears) based on FAF, Spectral Domain Optical Coherence Tomography (SD-OCT) imaging, intravenous fluorescein angiography (IVFA) and color fundus photo as assessed by the Central Reading Center.
* Spherical equivalent of -8.00 diopters (D) myopia or higher in the study eye.
* Uncontrolled glaucoma in the study eye (Intraocular pressure [IOP] >25 mmHg despite treatment with anti- glaucoma medication) or history of neovascular glaucoma.
* History of glaucoma filtration surgery, minimally-invasive glaucoma surgery involving an implant, or vitrectomy surgery, or other procedure in the study eye that could affect drug distribution and/or clearance.
* Any current or prior ocular disease, other than geographic atrophy, that in the opinion of the Investigator could interfere with the conduct of the study including, but not limited to, insufficient pupil dilation, retinal or optic nerve disease, media opacity, or aphakia in the study eye.
* History of any prior IVT treatment for any indication in the study eye.
* Any prior treatment for AMD in the study eye (for example, surgical, radiation, thermotherapeutic, or laser intervention), except oral supplements or minerals.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2021-02-26 (Actual); Primary Completion 2023-03-28 (Actual); Study Completion 2023-09-13 (Actual)

PRIMARY OUTCOMES:
GA lesion growth rate | Baseline to Month 12
  Change in GA lesion area as assessed by fundus autofluorescence (FAF)

SECONDARY OUTCOMES:
Safety: Participants with treatment-emergent adverse events (TEAEs) | Baseline to Month 18
  Number of participants with TEAEs
Best corrected visual acuity (BCVA) | Baseline to Month 18
  Change from baseline in BCVA as assessed by the Early Treatment Diabetic Retinopathy Study (ETDRS) test chart
Low-luminance BCVA (LL-BCVA) | Baseline to Month 18
  Change from baseline in LL-BCVA
Low-luminance visual acuity deficit (LL-VD) | Baseline to Month 18
  Change from baseline in LL-VD

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Annexon, Inc.
Locations (53):
- United States (45):
  - Site 5, Phoenix, Arizona
  - Site 31, Bakersfield, California
  - Site 2, Beverly Hills, California
  - Site 19, Mountain View, California
  - Site 23, Pasadena, California
  - Site 37, Poway, California
  - Site 17, Sacramento, California
  - Site 18, Santa Ana, California
  - Site 33, Walnut Creek, California
  - Site 39, Waterford, Connecticut
  - Site 12, Fort Myers, Florida
  - Site 53, Jacksonville, Florida
  - Site 26, Pensacola, Florida
  - Site 16, Pinellas Park, Florida
  - Site 43, Sarasota, Florida
  - Site 28, St. Petersburg, Florida
  - Site 6, Winter Haven, Florida
  - Site 42, Augusta, Georgia
  - Site 11, Lexington, Kentucky
  - Site 1, Hagerstown, Maryland
  - Site 41, Hagerstown, Maryland
  - Site 36, Boston, Massachusetts
  - Site 3, Springfield, Massachusetts
  - Site 29, Royal Oak, Michigan
  - Site 10, Reno, Nevada
  - Site 38, Bloomfield, New Jersey
  - Site 9, Cherry Hill, New Jersey
  - Site 30, Albuquerque, New Mexico
  - Site 20, Asheville, North Carolina
  - Site 52, Cleveland, Ohio
  - Site 13, Edmond, Oklahoma
  - Site 40, Eugene, Oregon
  - Site 27, Philadelphia, Pennsylvania
  - Site 15, Abilene, Texas
  - Site 4, Austin, Texas
  - Site 24, Bellaire, Texas
  - Site 34, Burleson, Texas
  - Site 21, Dallas, Texas
  - Site 32, Fort Worth, Texas
  - Site 22, Fort Worth, Texas
  - Site 35, Katy, Texas
  - Site 54, San Antonio, Texas
  - Site 8, San Antonio, Texas
  - Site 14, Charlottesville, Virginia
  - Site 25, Norfolk, Virginia
- Australia (6):
  - Site 49, Bondi Junction, New South Wales
  - Site 45, Brookvale, New South Wales
  - Site 46, Chatswood, New South Wales
  - Site 44, Sydney, New South Wales
  - Site 47, Sydney, New South Wales
  - Site 48, Adelaide, South Australia
- New Zealand (2):
  - Site 50, Christchurch
  - Site 51, Wellington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tzoumas N, Riding G, Williams MA, Steel DH. Complement inhibitors for age-related macular degeneration. Cochrane Database Syst Rev. 2023 Jun 14;6(6):CD009300. doi: 10.1002/14651858.CD009300.pub3. PMID 37314061